CLINICAL TRIAL: NCT04554030
Title: Impact of Immunotherapy in the Spermogram
Brief Title: Impact of Immunotherapy on the Sperm Count of Patients With Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, JOSE NICOLAS MINATTA, Principal investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 4019
Record Dates: First submitted 2020-01-02; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Sperm Count, Low
MeSH Terms: conditions — Oligospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Evaluate sperm count before and after immunotherapy — Evaluate sperm count before and after immunotherapy

SUMMARY:
Cancer is a public health problem. In recent years, oncology has been revolutionized with the advent of new treatments for different tumor models, mainly immunotherapy directed against cell cycle control points. Numerous inhibitory pathways are incorporated into the immune system to maintain tolerance and homeostasis, and these are collectively known as immunological checkpoints.

The main function of immunological checkpoints is to protect tissues from damage when the immune system is responding to pathogens and maintain tolerance to self antigens (ie, prevent autoimmunity). This is mainly achieved by down-regulation of T cell activation or effector functions. There is increasing evidence to show that a primary mechanism by which tumors evade the immune system is through the participation of immunological checkpoints. This has stimulated the development of many novel agents that modulate immunological checkpoints or other costimulatory receptors.

CTLA-4 is the first receptor of the checkpoint that is successfully selected as immunotherapy. Ipilimumab, an anti-CTLA-4 monoclonal antibody, was the first immunological checkpoint inhibitor to receive FDA approval for the treatment of advanced melanoma.

On the other hand, PD-1 is another receptor for the immune control point, and its ligands, the programmed cell death ligand 1 (PD-L1) and PD-L2, also resulted in important therapeutic advances in cancer immunotherapy.

Unlike CTLA-4, PD-1 is widely expressed and can be found in, in addition to T cells, in B cells and natural killer (NK) cells. The main function of PD-1 is to limit the activity of T cells in peripheral tissues during an inflammatory immune response.

The tumors can exploit this control point, expressing the ligand PD-L1 and generating that the cytotoxic T lymphocytes and the NK cells are anergic and incapable of killing. This up-regulation mechanism of PD-L1 is known in tumors such as melanoma, lung and ovary. Several monoclonal antibodies directed to PD-1 have already received approvals for their clinical use as Nivolumab and Pembrolizumab.

DETAILED DESCRIPTION:
The toxic effect of cytostatics (chemotherapy) at the gonadal level is known, but the effect that anti PD-1 immunotherapy can have on the spermogram of oncological patients at the level of the blood-testicular barrier, endocrine axis, among others, is not known. The proinflammatory mechanisms of immunotherapy could incur in damage evidenced as quali-quantitative alterations of the spermogram.

Primary end point:

To evaluate the difference in spermogram (counting, functionality, vitality, mobility) before and after treatment with anti-PD1 immunotherapy first line of oncological treatment of adult patients

Secondary end point:

Evaluate the association adjusted for nutrition, endocrine disorders. Evaluate modifications in the sexual functionality of patients through validated sexuality questionnaires before and during treatment.

In the absence of information, according to the results obtained, cryopreservation prior to the start of treatment could be taken into consideration.

Design: Observational prospective cohort with a single group. With start of follow-up from the oncological diagnosis of patients who are in the process of starting treatment with immunotherapy, checkpoint inhibitors in first line setting. The spermogram samples will be performed: 2 baseline before the start of the drug and +/- 5 days of the start of the treatment, separated by at least 2 weeks. Subsequent samples will be taken 3, 6 and 12 months after the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of cancer with indication for treatment with immunotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men on treatment with immunotherapy with check point inhibitors for cancer disease.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the difference in the spermogram before and after immunotherapy exposure | through study completion, an average of 1 year
  To determine differences in sperm count before and after exposure to immunotherapy. Count measured in cells / mm3

CONTACTS AND LOCATIONS:
Locations (1):
- Nicolas Minatta, Capital Federal, Argentina